CLINICAL TRIAL: NCT02677935
Title: Impact of Peer Education Program on Headache Disorders in Rural Communities, India: a Quasi-experimental Study
Brief Title: Impact of Peer Education Program on Headache Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Kaithal Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nmp/22182
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Headache Disorder
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): community support program
  Interventions: Other: Community education programs

INTERVENTIONS:
Other: Community education programs

SUMMARY:
Worldwide, headache disorders are among the most common medical conditions. Many people with headache need not experience further pain if the diagnosis and treatment are correct. Most patients do not have correct diagnosis and treatment. This study tested a model for treatment of people with headache disorders at primary health-care level in rural areas of Haryana, India.

ELIGIBILITY:
Inclusion Criteria:

* All residents of the Region Kaithal (haryana) may apply for recruitment
* Primary headache disorders including tension type headache, migraine

Exclusion Criteria:

* Planning to move the area
* Refused to consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Reduction in number of days per month with headache after 12 months | From baseline to 12 months

SECONDARY OUTCOMES:
Reduction in number of days per month of over the counter drugs after 12 months | From Baseline to 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Rani, Principal Investigator — NMP Medical Research Institute; Neeraj Kumar, Principal Investigator — Kaithal Hospital; Ram Sharma, Study Director — NMP Medical Research Institute

IPD SHARING:
Plan to Share IPD: Yes